CLINICAL TRIAL: NCT02202382
Title: Effects of Korean Red Ginseng on Male Infertility
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pusan National University Hospital (Other)
Responsible Party: Principal Investigator, Hyun Jun Park, Professor, Pusan National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KGR study
Record Dates: First submitted 2014-07-22; First posted 2014-07-29 (Estimated); Last update posted 2014-07-31 (Estimated); Status verified 2014-07

CONDITIONS: Male Infertility
MeSH Terms: conditions — Infertility, Male | interventions — Asian ginseng

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- non-V + P group (Placebo Comparator): no surgery and placebo (12 weeks)
  Interventions: Drug: Placebo
- V + P group (Active Comparator): Surgery with placebo (12 weeks)
  Interventions: Drug: Placebo; Procedure: Varicocelectomy
- non-V + KRG group (Active Comparator): no surgery with KRG (korean red ginseng, 1.5 gm daily 12weeks)
  Interventions: Drug: Korean Red Ginseng, Varicocelectomy
- V + KRG group (Experimental): Surgery with KRG (1.5 gm daily 12weeks)
  Interventions: Drug: Korean Red Ginseng, Varicocelectomy; Procedure: Varicocelectomy

INTERVENTIONS:
Drug: Korean Red Ginseng, Varicocelectomy
  Arms: V + KRG group; non-V + KRG group
Drug: Placebo — Placebo were provided by Korean Ginseng Corporation (Daejeon, Korea). The placebo capsules were identical in shape, color, and taste.
  Arms: V + P group; non-V + P group
Procedure: Varicocelectomy — Surgical microscope-assisted varicocelectomy using the subinguinal approach was conducted by a single surgeon.
  Arms: V + KRG group; V + P group

SUMMARY:
Objective: Several in vitro studies report positive effects of ginseng on spermatogenesis. However, no controlled human clinical study of the effect of Korean red ginseng (KRG) on spermatogenesis has been performed. This study was performed to investigate the effects of KRG on semen parameters in male infertility patients in a randomized, double-blind, placebo-controlled study. Methods: A total of 80 male infertility patients with varicocele were recruited from April 2011 to February 2012. The subjects were then divided into the following four groups: non-V + P group, placebo; V + P group, placebo and varicocelectomy; non-V + KRG group, 1.5-g KRG daily; V + KGR group, 1.5-g KRG daily and varicocelectomy. Semen analysis was performed and hormonal levels were measured in each treatment arm after 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients should be males, 25 - 45 years of age
* Complained of infertility for at least 12 months
* No history of surgical or medical treatments for infertility
* Increased retrograde flow in the internal spermatic vein with venous diameter > 3 mm during the Valsalva maneuver on scrotal ultrasonography was used as an indicator of varicocele.13 Varicocele was graded according to the criteria presented by Lyon et al.14: grade I, palpable only with the Valsalva maneuver; Grade II, palpable without the Valsalva maneuver; Grade III, visible from a distance.

Exclusion Criteria:

* The exclusion criteria were as follows:
* A history of vasectomy or obstructive azoospermia
* Chromosomal abnormalities
* Hypogonadism or pituitary abnormalities
* Anatomical abnormality of the genitals
* Significant hepatopathy (liver enzymes elevated 2 - 3-fold higher than the normal range)
* Renal insufficiency (serum creatinine level > 2.5 mg/dL)
* Medical treatment for infertility during the past 4 weeks

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2011-04; Primary Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Sperm concentration | When 12 week treatments were finished in all treatment arms, semen analysis and determination of hormonal levels were performed after 2 weeks of washout period
  Primary outcome measure according to World Health Organization (WHO) methodologies (4th edition)
Sperm motility | When 12 week treatments were finished in all treatment arms, semen analysis and determination of hormonal levels were performed after 2 weeks of washout period
  Primary outcome measure according to World Health Organization (WHO) methodologies (4th edition)
Sperm morphology | When 12 week treatments were finished in all treatment arms, semen analysis and determination of hormonal levels were performed after 2 weeks of washout period
  Primary outcome measure according to World Health Organization (WHO) methodologies (4th edition)
Sperm viability | When 12 week treatments were finished in all treatment arms, semen analysis and determination of hormonal levels were performed after 2 weeks of washout period
  Primary outcome measure according to World Health Organization (WHO) methodologies (4th edition)

SECONDARY OUTCOMES:
Serum concentrations of FSH | The hormonal status of all patients was recorded at the initial screening visit and post-treatment. (baseline and 12weeks after treatment)
  Serum hormonal levels were quantified by chemiluminescence assays
Serum concentrations of LH | The hormonal status of all patients was recorded at the initial screening visit and post-treatment. (baseline and 12weeks after treatment)
  Serum hormonal levels were quantified by chemiluminescence assays
Serum concentrations of testosterone | The hormonal status of all patients was recorded at the initial screening visit and post-treatment. (baseline and 12weeks after treatment)
  Serum hormonal levels were quantified by radioimmunoassay

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Urology, Pusan National University Hospital, Busan, South Korea